CLINICAL TRIAL: NCT00994656
Title: Is the Pleth Variability Index (PVI) a Useful Surrogate for Pulse Pressure Variations (PPV) in a Pediatric Population Undergoing Spine Fusion?
Brief Title: Is Pleth Variability Index (PVI) a Surrogate for Pulse Pressure Variations (PPV) in Pediatric Spine Fusion (SF) Surgery?
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Jeffrey Feldman, MD, The Children's Hospital of Philadelphia
Other Study IDs: 09-007194
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Scoliosis; Spinal Fusion
Keywords: invasive procedures; hypovolemia
MeSH Terms: conditions — Scoliosis; Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- posterior spinal fusion subject: Subject will have a history of either idiopathic or neuromuscular scoliosis who is now scheduled to have a posterior spinal fusion.
  Interventions: Device: Masimo multi-wavelength pulse co-oximeter

INTERVENTIONS:
Device: Masimo multi-wavelength pulse co-oximeter — Subjects will have a finger probe that will measure the pleth variability index. They will also have an arterial line (as standard of care) from which arterial pulse tracings will be obtained.
  Other Names: Masimo Rainbow Set; pulse co-oximeter

SUMMARY:
Spine fusion is an involved procedure during which patients are at risk for significant intra-operative blood loss.This study will compare 2 ways of determining fluid status and response to fluid administration. One way is to measure the changes in the arterial wave form from the special IV that is usually placed in an artery (PPV). The second way is to use a non-invasive method of a finger probe that measures changes in the plethysmogram or the pleth variability index (PVI). No actual patient treatments will be based on these values during surgery.

DETAILED DESCRIPTION:
Spine fusion is an involved procedure during which patients are at risk for significant intra-operative blood loss. The resulting hypovolemia increases the fluctuations in arterial pressure associated with positive pressure ventilation. These respiratory induced arterial pressure variations (RIAPV) appear as cyclical peaks and troughs on the arterial waveform.

Different approaches have been used to quantify the RIAPV. One such approach has been to measure the pulse pressure variation (PPV), using invasive arterial monitoring. In previous studies, PPV has been shown to be a good indicator of fluid responsiveness intra-operatively, but this has not been specifically evaluated in patients undergoing spine fusion. This patient population is of particular interest because of their underlying scoliosis as well as their prone position during the operation. These two variables could potentially alter lung-thorax mechanics in a manner which may influence RIAPV, which is specifically determined by the interaction between intrathoracic pressure and venous filling of the heart. A second approach to quantifying RIAPV relies on non invasive technology initially developed by the Masimo Corporation for pulse oximetry. This parameter has been coined pleth variability index (PVI), as it specifically quantifies real time changes in the plethysmogram associated with respiration. PVI, which is based on arterial blood volume changes, is therefore analogous to PPV, which is derived from changes in arterial pressure. To date PVI has only been evaluated in adult patients undergoing cardiac surgery and the data suggest that it may be a useful indicator of fluid responsiveness.

Given the non-invasive and continuous nature of PVI, it is appealing for potential use as a bedside monitor to guide fluid resuscitation. However, photoplethysmography is known to be sensitive to noise due to motion, light and electrical interference. Furthermore, PVI is based upon a degree of quantitative evaluation of the photoplethysmogram that is the first of its kind. For these reasons, it is important to understand the limits of agreement between PVI and PPV before we can accept PVI as a non-invasive surrogate measurement. This study intends to evaluate PVI by analyzing it in relation to PPV. More specifically, paired measurements of PPV and PVI will be compared to determine the limits of agreement between the two parameters in patients undergoing spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 8 to 18 years inclusive.
* History of idiopathic or neuromuscular scoliosis.
* Scheduled for posterior spinal fusion.
* Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

* Inability to understand or read English to provide consent.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be selected from those having posterior spinal fusion surgery at The Children's Hospital of Philadelphia.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Feldman, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States